CLINICAL TRIAL: NCT01288742
Title: A Phase I, 2-panel, Open-label, Randomized, Crossover Trial in Healthy Subjects to Investigate the Pharmacokinetic Interaction Between TMC435 and Transporter Substrates, Digoxin and Rosuvastatin
Brief Title: TMC435-TiDP16-C108 - A Study in Healthy Volunteers Investigating the Pharmacokinetic Interaction Between TMC435 and Digoxin and Between TMC435 and Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR017770; TMC435-TiDP16-C108
Record Dates: First submitted 2011-01-20; First posted 2011-02-02 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Hepatitis C Virus
Keywords: TMC435-TiDP16-C108; TMC435-C108; TMC435; HPC; HCV; Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Rosuvastatin Calcium; Simeprevir; Digoxin

ARMS (5):
- 001 (Experimental): TMC435 One 150-mg capsule once daily for 7 days (Trts B and D).
  Interventions: Drug: TMC435
- 002 (Experimental): Digoxin One 0.25-mg tablet for 1 day (Trt A)
  Interventions: Drug: Digoxin
- 003 (Experimental): Digoxin One 0.25-mg tablet together with 1 capsule of TMC435 (150 mg) on Day 7 of Trt B.
  Interventions: Drug: Digoxin
- 004 (Experimental): Rosuvastatin One 10-mg tablet for 1 day (Trt C).
  Interventions: Drug: Rosuvastatin
- 005 (Experimental): Rosuvastatin One 10-mg tablet together with 1 capsule of TMC435 (150 mg) on Day 7 of Trt D.
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — One 10-mg tablet for 1 day (Trt C).
  Arms: 004
Drug: Rosuvastatin — One 10-mg tablet together with 1 capsule of TMC435 (150 mg) on Day 7 of Trt D.
  Arms: 005
Drug: TMC435 — One 150-mg capsule once daily for 7 days (Trts B and D).
  Arms: 001
Drug: Digoxin — One 0.25-mg tablet together with 1 capsule of TMC435 (150 mg) on Day 7 of Trt B.
  Arms: 003
Drug: Digoxin — One 0.25-mg tablet for 1 day (Trt A)
  Arms: 002

SUMMARY:
The purpose of this study is to investigate the effect of steady-state concentrations of TMC435 on the single-dose pharmacokinetics of digoxin or rosuvastatin , and the effect of a single dose of digoxin or rosuvastatin on the steady-state pharmacokinetics of TMC435. Steady state is a term that means that the drug has been given long enough so that the plasma concentrations will remain the same with each subsequent dose. TMC435 is being investigated for the treatment of chronic hepatitis C virus (HCV) infection. Pharmacokinetics (PK) means how the drug is absorbed into the bloodstream, distributed in the body, and eliminated from the body.

DETAILED DESCRIPTION:
TMC435 is being investigated for treatment of chronic hepatitis C virus (HCV) infection, in combination with Peg-IFN (pegylated interferon) and RBV (ribavirin). Digoxin and rosuvastatin are expressed in the liver and intestine and mediate the transport of drugs out of the blood circulation. The result of this study will provide dosing recommendations for TMC435 and for digoxin, rosuvastatin, or other substrates using the same drug transporter molecules, when being coadministered. This is a Phase I, open-label (both participant and investigator know the name of the medication given at certain moment), randomized (sequence of treatment with study medications is assigned by chance), crossover trial in 32 healthy volunteers to investigate the pharmacokinetic interaction between TMC435, at steady state, and digoxin or rosuvastatin at a single dose. The volunteers will be allocated to one of two panels. In Panel 1, volunteers will receive two treatments (Trts A and B) in a randomized order. Volunteers will receive digoxin 0.25 mg once daily for 1 day (Trt A) and TMC435 150 mg once daily for 7 days (Trt B) and 0.25 mg digoxin once daily for 1 day (Trt B). In Panel 2, volunteers will receive two treatments (Trts C and D) in a randomized order. Volunteers will receive rosuvastatin 10 mg once daily for 1 day (Trt C) and TMC435 150 mg once daily for 7 days (Trt D) and rosuvastatin 10 mg once daily for 1 day (Trt D). In both panels, there will be a washout period (a period when no study drug will be taken, in order to have all the medication eliminated from the body before starting a new treatment) of at least 14 days between last intake of the study medication in one session and the first intake of study medication in the subsequent session. Pharmacokinetic profiles of all three compounds will be determined through blood samples taken at regular intervals during the study. Safety and tolerability will be assessed during the study period and during follow up. Blood and urine samples, electrocardiogram (ECG) and vital signs (blood pressure and heart rate) will be taken at screening, before medication intake on Day -1 or Day 1 (Trts A, B, C, and D), on Day 2 (Trts A and C), before medication intake and 6 hours postdose (only vital signs and ECG) on Day 7 (Trts B and D), on Day 8 (Trts B and D) and at the 2 follow up visits at 1 week and 4-5 weeks after last dose of study medication in the last session. A physical examination will be performed at screening, on Day -1 (= day before first medication intake in each session for both panels) and on Day 2 in Trts A and C, on Day -1 and on Day 8 of Trts B and D and during the 2 follow-up visits. Each volunteer is part of one panel and follows 2 treatment (Trt) periods, which are a minimum 14 days apart from each other. Trt period for Trts A and C - 5 days; Trt period for Trts B and D - 11 days. Trt A and B = Panel 1, Trt C and D = Panel 2. A single, oral dose of digoxin (0.25 mg) or rosuvastatin (10 mg) to be given in Trt A or Trt C, respectively. Multiple doses of TMC435 (150 mg) for 7 days to be given in TrtB and D, with a single dose of digoxin or rosuvastatin on Day7, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker or not having chewed tobacco for at least 6 months
* Body Mass Index of 18.0 to 30.0 kg/m2
* Healthy based on a medical evaluation including medical history, physical examination, blood tests, vital signs, and electrocardiogram

Exclusion Criteria:

* Infection with hepatitis A, B or C virus
* Infection with the human immunodeficiency virus (HIV)
* History of, or any current medical condition which could impact the safety of the participant in the study
* Having previously participated in a multiple-dose trial with TMC435
* Having previously participated in more than 3 single-dose trials with TMC435
* History of rhabdomyolysis or other muscle abnormalities upon statin intake (Panel 2).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change in absorption of TMC435 following co-administration with Digoxin (Panel 1). | Measured on Days 1, 5-11 (Trt B). Reference for TMC435 is from historical data.
Change in absorption of Digoxin following co-administration with TMC435 (Panel 1). | Measured on Day 7-11 (Trt B). Reference for Digoxin is on Day 1-5 of Trt A.
Change in absorption of TMC435 following co-administration with rosuvastatin (Panel 2). | Measured on Day 1, 5-11 (Trt D). Reference for TMC435 are historical data.
Change in absorption of rosuvastatin following co-administration with TMC435 (Panel 2). | Measured on Day 7-11 (Trt D). Reference for rosuvastatin is on Days 1-5 of Trt C.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability - TMC435 and Digoxin | 51 to 56 days (until and including last safety follow-up visit) for Panel 1
Number of participants with adverse events as a measure of safety and tolerability - TMC435 and rosuvastatin | 51 to 56 days (until and including last safety follow-up visit) for Panel 2

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited